CLINICAL TRIAL: NCT05126290
Title: CTNNA1 Familial Expansion (CAFÉ) Study
Brief Title: CTNNA1 Familial Expansion Study
Acronym: CAFÉ
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Bryson Katona, Assistant Professor of Medicine, Director - Gastrointestinal Cancer Genetics Program, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 21220; 844070 (Other: UPENN IRB)
Record Dates: First submitted 2021-11-02; First posted 2021-11-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cancer Gene Mutation; Gastric Cancer; Breast Cancer
Keywords: CTNNA1; Hereditary diffuse gastric cancer; Gastric cancer; Breast cancer
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of personal and family history from CAFÉ Study participants — Personal medical and genetic history, as well as relevant information about family history, will be collected from participants in the CAFÉ Study through an online data entry system

SUMMARY:
The goal of the CAFÉ Study is to determine the cancer risks associated with germline CTNNA1 loss-of-function variants.

DETAILED DESCRIPTION:
The CAFÉ Study aims to determine the degree to which loss-of-function variants in the CTNNA1 gene are associated with hereditary cancers, including gastric cancer, breast cancer, as well as other cancers that may be associated with this gene. By obtaining personal and family history information from individuals who carry a CTNNA1 loss-of-function variant and their family members, this study will aim to better define CTNNA1 associated cancer risks and determine whether there is a genotype/phenotype correlation for CTNNA1 loss-of-function variants. This information will be important for the future cancer risk management of individuals who carry a CTNNA1 loss-of-function variant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Participants must be carrier, or a first degree relative of a carrier, of a CTNNA1 loss-of-function variant defined as: a variant predicted to lead to protein truncation (nonsense and frameshift variants), a large deletion of one or more exons, or a consensus splice site variant predicted to disrupt splicing in CTNNA1. CTNNA1 loss-of-function variants do not need to be classified as pathogenic or likely pathogenic to be included.
* Participants must be able to understand and read English
* Participants must be able to provide informed verbal or written consent

Exclusion Criteria:

* Less than 18 years of age
* Individuals who do not carry a CTNNA1 loss-of-function variant and are not a first degree relative of a CTNNA1 loss-of-function variant carrier.
* Individuals who cannot speak and read English
* Major psychiatric illness or cognitive impairment that in the judgement of the study investigators or study staff would preclude study participation
* Unable to comply with the study procedures as determined by the study investigators or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CAFÉ Study will recruit individuals who carry a germline CTNNA1 loss-of-function variant as well as first degree relatives of germline CTNNA1 loss-of-function variant carriers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of cancer amongst carriers of CTNNA1 loss-of-function variants | Through study completion, which will average 1 year
  After collecting personal and family cancer history from enrolled participants, family pedigrees will be utilized to calculate cancer risk estimates for for CTNNA1 loss-of-function variant carriers including gastric cancer risk, breast cancer risk, as well as risk of other cancers currently not known to be associated with CTNNA1 variants gene.
Number of CTNNA1 genotypes associated with a cancer phenotype | Through study completion, which will average 1 year
  Using collected family pedigrees from enrolled participants, we will correlate estimated cancer risk for CTNNA1 loss-of-function variant carriers with their CTNNA1 genotype, to determine if there is a significant genotype-phenotype correlation observed.

CONTACTS AND LOCATIONS:
Overall Officials: Bryson W Katona, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark DF, Michalski ST, Tondon R, Nehoray B, Ebrahimzadeh J, Hughes SK, Soper ER, Domchek SM, Rustgi AK, Pineda-Alvarez D, Anderson MJ, Katona BW. Loss-of-function variants in CTNNA1 detected on multigene panel testing in individuals with gastric or breast cancer. Genet Med. 2020 May;22(5):840-846. doi: 10.1038/s41436-020-0753-1. Epub 2020 Feb 13. PMID 32051609
- See also: Study website — http://www.pennmedicine.org/CAFEStudy